CLINICAL TRIAL: NCT06604013
Title: Class III Obesity and Periodontitis: Gingival Crevicular Fluid of Adiponectin and Resistin As Predictable Implement in Staging and Grading System and Effects of Periodontal Therapy
Brief Title: Gingival Crevicular Fluid of Adiponectin and Resistin As Predictable Implement in Staging and Grading System of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asem Mohammed Kamel Ali, lecturer, Al-Azhar University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Obesity and Periodontitis
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Periodontal Diseases; Obesity, Morbid
Keywords: resistin, adiponectin, periodontitis Grading, periodontal therapy
MeSH Terms: conditions — Periodontal Diseases; Obesity, Morbid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- mild periodontitis (first stage, grade B) (Active Comparator): mild periodontitis (first stage, grade B) manifesting CAL ≥ 1-2 mm, in corporation with percentage of bone loss level divided by age was 0.25-1% very year. patients received non-surgical full-mouth periodontal therapy without using adjunct disinfectants.
  Interventions: Procedure: non-surgical full-mouth periodontal therapy without using adjunct disinfectants; Diagnostic Test: GCF level of adiponectin and resistin
- moderate periodontitis (second stage, grade B) (Active Comparator): moderate periodontitis (second stage, grade B) manifesting CAL ≥ 3-4mm in corporation with percentage of bone loss level divided by age was 0.25-1% very year. patients received non-surgical full-mouth periodontal therapy without using adjunct disinfectants.
  Interventions: Procedure: non-surgical full-mouth periodontal therapy without using adjunct disinfectants; Diagnostic Test: GCF level of adiponectin and resistin
- severe periodontitis (third stage, grade B) (Active Comparator): severe periodontitis (third stage, grade B) manifesting CAL ≥ 5mm , in corporation with BoP increased than (30%), percentage of bone loss level divided by age was 0.25-1% very year. patients received non-surgical full-mouth periodontal therapy without using adjunct disinfectants
  Interventions: Procedure: non-surgical full-mouth periodontal therapy without using adjunct disinfectants; Diagnostic Test: GCF level of adiponectin and resistin
- very severe periodontitis (forth stage, grade C) (Active Comparator): very severe periodontitis (forth stage, grade C) manifesting CAL ≥ 5mm in corporation of percentage of bone loss level divided by age more than 1% very year. patients received non-surgical full-mouth periodontal therapy without using adjunct disinfectants
  Interventions: Procedure: non-surgical full-mouth periodontal therapy without using adjunct disinfectants; Diagnostic Test: GCF level of adiponectin and resistin

INTERVENTIONS:
Procedure: non-surgical full-mouth periodontal therapy without using adjunct disinfectants — Supragingival scaling was performed by Ultrasonic Scaler and manual scaling by sickle scaler . Subgingival scaling and root planing were accomplished with either universal or area specific Gracey curettes
Diagnostic Test: GCF level of adiponectin and resistin — Gingival crevicular fluid (GCF) samples were gathered and relocated in phosphate buffer saline inside Eppendorf tube then t they were manipulated by commercially available enzyme-linked immuno-sorbent assay

SUMMARY:
The goal of this clinical trial is to evaluate the relationship between obesity and gingival crevicular fluid resistin and adiponectin in periodontitis patients as well as assess the effect of non-surgical periodontal therapy on their levels using ELISA in obese individuals. Researchers will compare different stages of periodontitis to see if degrees of inflammation and periodontal therapy related obesity

ELIGIBILITY:
Inclusion Criteria:

* obese persons with Body Mass Index (BMI) more than 40 and suffering from periodontitis

Exclusion Criteria:

* Patients receiving either antibiotics or non-steroidal anti- inflammatory at least 3 months prior to samples collection.
* Patients subjected to previous periodontal therapy 6 months before sampling. Patients with systemic or local inflammatory conditions other than periodontal disease.
* Neither lactating nor pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
adiponectin level in gingival crevicular fluid | From enrollment to the end of treatment results assessment at 12 weeks
resistin level in gingival crevicular fluid | From enrollment to the end of treatment results assessment at 12 weeks

SECONDARY OUTCOMES:
O'Leary Plaque score | From enrollment to the end of treatment results assessment at 12 weeks
bleeding on probing percentage (BoP) | From enrollment to the end of treatment results assessment at 12 weeks
clinical attachment level (CAL) | From enrollment to the end of treatment results assessment at 12 weeks
probing pocket depth | From enrollment to the end of treatment results assessment at 12 weeks

OTHER OUTCOMES:
Body Mass Index (BMI) | From enrollment time only
glycated hemoglobin (HbA1c) | From enrollment time only

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa Mohammed Badr, associate professor, Study Director — Faculty of dental medicine Al-Azhar university Assiut Branch; Asem Mohammed kamel, lecturer, Study Director — Faculty of dental medicine Al-Azhar university Assiut Branch
Locations (1):
- Faculty of Dental Medicine, Al-Azhar University Assiut Branch, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kusminski CM, McTernan PG, Kumar S. Role of resistin in obesity, insulin resistance and Type II diabetes. Clin Sci (Lond). 2005 Sep;109(3):243-56. doi: 10.1042/CS20050078. PMID 16104844
- [Background] Filkova M, Haluzik M, Gay S, Senolt L. The role of resistin as a regulator of inflammation: Implications for various human pathologies. Clin Immunol. 2009 Nov;133(2):157-70. doi: 10.1016/j.clim.2009.07.013. Epub 2009 Sep 8. PMID 19740705
- [Background] Cugini MA, Haffajee AD, Smith C, Kent RL Jr, Socransky SS. The effect of scaling and root planing on the clinical and microbiological parameters of periodontal diseases: 12-month results. J Clin Periodontol. 2000 Jan;27(1):30-6. doi: 10.1034/j.1600-051x.2000.027001030.x. PMID 10674959